CLINICAL TRIAL: NCT05945108
Title: Brazilian Reality of Urinary Bladder Cancers - BRA-BLADDER: Multicenter Retrospective Study (Real World Evidence - RWE)
Brief Title: Brazilian Reality of Urinary Bladder Cancers - BRA-BLADDER
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: D133HR00023
Record Dates: First submitted 2023-06-22; First posted 2023-07-14 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Urothelial Carcinoma; Non Muscle Invasive Bladder Cancer; Muscle-invasive Bladder Cancer
Keywords: Bladder Cancer, RWE
MeSH Terms: conditions — Carcinoma, Transitional Cell; Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-muscle-invasive bladder cancer or Muscle-invasive bladder cancer: Defined as:
  * T1 tumor and/or high-grade lesion (G3) and/or presence of CIS (Carcinoma in situ).
  * Multifocal relapsed tumor and with at least one large lesion (diameter ≥ 3 cm);
  Or:
  -Diagnosis of early muscle-invasive urothelial bladder carcinoma.

SUMMARY:
A national, multicenter, non-randomized, retrospective, observational study (Real-World Evidence-RWE) aimed at analyzing clinical presentation profiles and demographic characteristics of patients with early urothelial bladder cancer (high-risk non-muscle invasive and localized muscle-invasive) treated with standard therapies in national cancer treatment reference centers within the last 6 years (between 2017 and 2022).

DETAILED DESCRIPTION:
Urothelial carcinoma has several histological types, extensive genetic diversity and a wide array of risk factors related to disease development. Moreover, the treatment effectiveness may be widely impacted by factors such as age, previous comorbidities, socio-economic factors, late diagnosis and access to treatment. In the last decade, the treatment profile has evolved worldwide with the incorporation of new technologies, however, there is no data on Brazilian reality in this period. In a continent-sized country and such heterogeneous health services as Brazil, preparing such knowledge becomes more important and challenging. This paper proposed to describe early urothelial carcinoma presentation pattern and treatment in Brazilian population (high-risk non-muscle-invasive and localized muscle-invasive) in several sites spread throughout the national territory. Thus, data will be generated to provide a more appropriate understanding of the current landscape and, consequently, the better design of public policies to face this disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old;
* Diagnosis of high-risk non-muscle invasive urothelial carcinoma, defined as:
* T1 tumor and/or high-grade lesion (G3) and/or presence of CIS.
* Multifocal relapsed tumor and with at least one large lesion (diameter ≥ 3 cm);
* Diagnosis of early muscle-invasive urothelial bladder carcinoma (cT2, cT3 or cT4a N0);
* Consent to participate in the study.

Exclusion Criteria:

* Low-risk non-muscle invasive urothelial carcinoma (single lesion, pTa and low-grade);
* Locally advanced muscle-invasive urothelial carcinoma (suspected lymph node impairment in staging imaging tests) or metastatic at diagnosis;
* Bladder carcinoma with non-urothelial histology (adenocarcinoma, squamous-cell carcinoma or small cell carcinoma);

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects to be enrolled are those with early urothelial carcinoma (high-risk non-muscle invasive and localized muscle-invasive), who meet the eligibility criteria and have been treated and followed in study participating sites within the last 6 years (period from 2017 to 2022).
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-04-18 (Actual)

PRIMARY OUTCOMES:
Clinical staging | At first diagnosis and over 6 years (Time of retrospective observational analysis of the study)
  Description of the characteristics of the lesions at the initial diagnosis, performed by histopathology and imaging exams.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Maluf, MD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (5):
- Brazil (5):
  - Research Site, Belo Horizonte
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, Salvador
  - Research Site, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133HR00023&attachmentIdentifier=a918b067-0f84-4dc9-9d2e-7d6ea5dee72b&fileName=Clinical_Study_Report_(CSR)_Synopsis,_PantumorBladder.pdf&versionIdentifier=